CLINICAL TRIAL: NCT01654263
Title: A Phase IIb, Open-Label, Dose-Ranging Study of 13-Valent Pneumococcal Conjugate Vaccine in Adults 55 Through 74 Years of Age Previously Vaccinated With 23-Valent Pneumococcal Polysaccharide Vaccine
Brief Title: A Phase IIb, Open-Label, Dose Ranging Study of 13-Valent Pneumococcal Conjugate Vaccine in Adults 55 Through 74 Years of Age Previously Vaccinated With 23-Valent Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 11-0034; HHSN272201300018I
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2016-04-15

CONDITIONS: Pneumococcal Infection
Keywords: 13-valent; 23-valent; elderly; parent protocol; Pneumococcal infections; vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; CRM197 (non-toxic variant of diphtheria toxin)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group IA: Pneumococcal vaccine-naive, age 55 - 64 (Experimental): Open- label, 13-valent pneumococcal conjugate vaccine (PCV13) given as 0.5 mL intramuscular (IM) injection to 147 subjects vaccine-naive adults
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]
- Group IB: Pneumococcal vaccine-naive, age 65 - 74 (Experimental): Open- label, PCV13 given as 0.5 mL IM injection to 147 subjects vaccine-naive adults
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]
- Group IIA: age 55 - 64, previous PPSV23 (Experimental): Open-label, randomized PCV13 given as a 0.5 mL IM injection to 147 subjects with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]
- Group IIAA: age 55 - 64, previous PPSV23 (Experimental): Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to 147 subjects with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]
- Group IIB: age 65 - 74, previous PPSV23 (Experimental): Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to 147 subjects with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]
- Group IIBB: age 65 - 74, previous PPSV23 (Experimental): Open-label, randomized PCV13 given as a 0.5 mL IM injection to 147 subjects with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]

INTERVENTIONS:
Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein] — Prevnar 13 (PCV13) 13-valent pneumococcal conjugate vaccine. All doses given on Day 0. Group IA and IB (open-label): 0.5 mL intramuscular (IM) injection; Group IIA (open-label, randomized): 0.5 mL IM injection; Group IIB (open-label, randomized): 0.5 mL IM injection in the right arm and 0.5 mL IM in the left arm.

SUMMARY:
The proposed phase IIb randomized, open label, dose ranging, safety and immunogenicity study will evaluate two different doses of 13-valent pneumococcal conjugate vaccine (PCV13) in two groups of participants (55 through 74 years of age). First group vaccine naïve participants will be open-label to receive a single injection of 0.5 mL PCV13. Second group of participant previously vaccinated with 23-valent pneumococcal polysaccharide vaccine (PPSV23) will be randomized 1:1 to receive two injections of 0.5 mL PCV13, one dose in each arm (Group IIA or Group IIB). Blood samples will be obtained at baseline, at one month and six months post-vaccination. The primary objectives are: to determine if two 0.5 mL doses of PCV13 are statistically significantly more immunogenic than a single 0.5 mL dose of PCV13 for at least some of the vaccine serotypes among participants 55 through 74 years of age previously vaccinated with PPSV23, as measured by serotype-specific OPA titers 28 days after study

DETAILED DESCRIPTION:
This is a phase IIb open-label immunogenicity and safety study to evaluate dosages of 0.5 mL and 1.0 mL (given as two 0.5 mL injections in separate arms) of PCV13 in adults 55 through 74 years of age previously vaccinated with PPSV23. The study will enroll two groups of participants. Group I participants will all receive an open-label dose of 0.5 mL PCV13 and will include 294 adults 55-74 years of age who have not previously received 23-valent pneumococcal polysaccharide vaccine (PPSV23). Group II will be randomized 1:1 to receive 0.5 mL PCV13 (Group IIA) or 0.5 mL PCV13 in the right arm and 0.5 mL PCV 13 in the left arm (Group IIB). Group II will include 588 adults 55 through 74 years of age who previously received a single dose of PPSV23 > /=3 years and < /=7 years prior to enrollment. Enrollment in both groups will be stratified by age group (55 through 64 years and 65 through 74 years).The study duration is approximately 18 months. The primary objectives are: to determine if two 0.5 mL doses of PCV13 are statistically significantly more immunogenic than a single 0.5 mL dose of PCV13 for at least some of the vaccine serotypes among participants 55 through 74 years of age previously vaccinated with PPSV23, as measured by serotype-specific OPA titers 28 days after study vaccination, and is non-inferior to 12 vaccine serotypes; and determine if two 0.5 mL doses of PCV13 administered to participants previously vaccinated with PPSV23 are non-inferior to a single dose of 0.5 mL of PCV13 administered to vaccine-naïve adults 55 through 74 years of age for the 12 vaccine serotypes, as measured by serotype-specific OPA titers 28 days after study vaccination. The secondary objectives of this study are to: determine if two x 0.5mL doses of PCV13 is statistically significantly more immunogenic than a single 0.5 mL dose of PCV13 for at least some of the vaccine serotypes among participants 55 through 74 years of age previously vaccinated with PPSV23, as measured by serotype-specific OPA titers 180 days after study vaccination, and is non-inferior to 12 vaccine serotypes; to determine if two x 0.5mL doses of PCV13 administered to participants previously vaccinated with PPSV23 is non-inferior to a single dose of 0.5 mL of PCV13 administered to vaccine-naïve adults 55 through 74 years of age for 12 vaccine serotypes, as measured by serotype-specific OPA titers 180 days after study vaccination. Parent protocol to sub-study 12-0031.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults 55 through 74 years of age at the time of enrollment who are able to provide informed consent. 2. For the pneumococcal vaccine-naïve group (Group I), no pneumococcal vaccine received prior to enrollment, as documented by participant report and review of available vaccine records. For the previously vaccinated group (Group II), documented vaccination with exactly one dose of PPSV23 administered >/=3 and </=7 years prior to enrollment and no other lifetime doses of PPSV23. (History of receipt or non-receipt of a pneumococcal vaccine may be presumptively ascertained by participant report but must be confirmed by review of primary source information, including but not limited to medical records, primary care or other provider report, and health department records. Medical records should be reviewed and/or primary care or other providers queried to identify pneumococcal vaccinations administered for a period of not less than 10 years prior to enrollment.) 3. Determined by medical history, targeted physical examination (if indicated), and clinical judgment to be eligible for the study. Subjects with preexisting stable disease, defined as disease not requiring significant change in therapy (A change in dose or therapy within a category (e.g., change from one nonsteroidal anti-inflammatory drug to another) is allowed. A change to a new therapy category (e.g. surgery or addition of a new pharmacological class) is only allowed if it is not caused by worsening disease.) or hospitalization for worsening disease 12 weeks prior to enrollment, are eligible. 4. Agree not to receive a live virus vaccine (for example, zoster vaccine) before the Day 28 (Visit 03) blood specimen collection and not to receive an inactivated vaccine (for example, inactivated influenza vaccine) within 14 days after enrollment. 5. The subject is able to understand and comply with the planned study procedures including being available for all study visits. 6. The subject has provided informed consent prior to any study procedures.

Exclusion Criteria:

1. Receipt of any PCV or investigational pneumococcal vaccine prior to enrollment. 2. Receipt of any inactivated vaccine within 14 days prior to enrollment or receipt of any live vaccine within 30 days prior to enrollment. 3. Receipt of an allergy desensitization injection within 14 days prior to enrollment or planned receipt of an allergy desensitization injection within 7 days following enrollment. 4. Receipt of a diphtheria toxoid containing vaccine (for example, tetanus and diphtheria toxoid [Td] or tetanus and diphtheria toxoid and acellular pertussis [TdaP] vaccine) within six months prior to enrollment. 5. Known or suspected immunodeficiency, receipt of cancer chemotherapy or radiation therapy within the preceding 36 months, or receiving treatment with immunosuppressive therapy, including systemic corticosteroids, e.g., for cancer, HIV or autoimmune disease. If any systemic (oral, parenteral) corticosteroids have been administered for treatment of acute illness within 30 days of vaccination, and any long term use (>2 weeks) in the 30 through 59 days before vaccination should be excluded. (Topical, intranasal, and inhaled corticosteroids are allowed.) 6. Serious chronic disorders including active or metastatic malignancy, hematologic malignancy, severe chronic obstructive pulmonary disease or clinically significant congestive heart failure, requirement for supplemental oxygen, end stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that in the opinion of the investigator precludes the subject's participation. 7. Known HIV, hepatitis B or hepatitis C infection. 8. Residence in a nursing home or other skilled nursing facility or requirement for skilled nursing care. An ambulatory subject who does not require skilled nursing care and is a resident of a retirement home or community is eligible for the trial. 9. Inability to provide informed consent or complete study activities, for example, due to dementia or other impairment. 10. Poor or missing eyesight, requiring third party support to read. 11. Receipt of any blood products, including immunoglobulin, within three months prior to enrollment. 12. Heart rate less than 40 bpm or greater than 120 bpm as measured at the enrollment visit and prior to vaccination. 13. Systolic blood pressure less than 90 mm Hg or greater than 170 mm Hg as measured at the enrollment visit and prior to vaccination. 14. Diastolic blood pressure greater than 110 mm Hg as measured at the enrollment visit and prior to vaccination. 15. For Group I, unable to receive a vaccination in the deltoid muscle of the right arm and unable to receive a vaccination in the deltoid muscle of the left arm because of insufficient muscle mass, need to avoid injections due to prior lymph node dissection or radiation, or other factor. For Group II, unable to receive a vaccination in the deltoid muscle of one or both arms because of insufficient muscle mass, need to avoid injections due to prior lymph node dissection or radiation, or other factor. 16. Currently on anticoagulant therapy (for example, warfarin, heparin [IV or SQ], or dabigatran) or a history of bleeding diathesis that would contraindicate intramuscular injection. (Aspirin, clopidogrel, dipyridamole, and nonsteroidal anti-inflammatory agents are allowed). 17. Known clinically significant allergic reaction to prior pneumococcal vaccination (for Group II participants) or to a component of PCV13 vaccine (PCV13 is latex free). 18. Current known abuse of alcohol or drug addiction that in the opinion of the Investigator may interfere with the subject's ability to comply with trial procedures. 19. Rec eipt of any other investigational vaccine or agent within one month before enrollment or intent to receive any other investigational vaccine or agent prior to the conclusion of the study. 20. Any medical condition that would, in the opinion of the investigator, place the participant at an unacceptable risk of an adverse event or interfere with the evaluation of the study objectives.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2015-08-21 (Actual); Study Completion 2015-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle - Vaccines and Infectious Diseases, Seattle, Washington

REFERENCES:
- [Derived] Jackson LA, El Sahly HM, George S, Winokur P, Edwards K, Brady RC, Rouphael N, Keitel WA, Mulligan MJ, Burton RL, Nakamura A, Ferreria J, Nahm MH. Randomized clinical trial of a single versus a double dose of 13-valent pneumococcal conjugate vaccine in adults 55 through 74 years of age previously vaccinated with 23-valent pneumococcal polysaccharide vaccine. Vaccine. 2018 Jan 29;36(5):606-614. doi: 10.1016/j.vaccine.2017.12.061. Epub 2017 Dec 24. PMID 29279281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and females, 55 through 74 years of age, recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 10OCT2012 and 03MAR2015.
Groups:
- IA: Pneumococcal Vaccine-naive, Age 55-64, Single Injection: Open- label, 13-valent pneumococcal conjugate vaccine (PCV13) given as 0.5 mL intramuscular (IM) injection to vaccine-naive adults ages 55-64.
- IB: Pneumococcal Vaccine-naive, Age 65-74, Single Injection: Open- label, 13-valent pneumococcal conjugate vaccine (PCV13) given as 0.5 mL intramuscular (IM) injection to vaccine-naive adults ages 65-74.
- IIA: Age 55-64, Previous PPSV23, Single Injection: Open-label, randomized PCV13 given as a 0.5 mL IM injection to adults ages 55-64 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- IIB: Age 65-74, Previous PPSV23, Single Injection: Open-label, randomized PCV13 given as a 0.5 mL IM injection to adults ages 65-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- IIAA: Age 55-64, Previous PPSV23, Two Injections: Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to adults ages 55-64 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- IIBB: Age 65 - 74, Previous PPSV23, Two Injections: Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to adults ages 65-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
Period: Overall Study
Arm/Group | IA: Pneumococcal Vaccine-naive, Age 55-64, Single Injection | IB: Pneumococcal Vaccine-naive, Age 65-74, Single Injection | IIA: Age 55-64, Previous PPSV23, Single Injection | IIB: Age 65-74, Previous PPSV23, Single Injection | IIAA: Age 55-64, Previous PPSV23, Two Injections | IIBB: Age 65 - 74, Previous PPSV23, Two Injections
Started | 164 | 147 | 139 | 145 | 140 | 149
Completed | 164 | 147 | 137 | 144 | 139 | 148
Not Completed | 0 | 0 | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants are included in the baseline analysis population.
Groups:
- IIBB: Age 65-74, Previous PPSV23, Two Injections: Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to adults ages 65-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- Total: Total of all reporting groups
Arm/Group | IA: Pneumococcal Vaccine-naive, Age 55-64, Single Injection | IB: Pneumococcal Vaccine-naive, Age 65-74, Single Injection | IIA: Age 55-64, Previous PPSV23, Single Injection | IIB: Age 65-74, Previous PPSV23, Single Injection | IIAA: Age 55-64, Previous PPSV23, Two Injections | IIBB: Age 65-74, Previous PPSV23, Two Injections | Total
Number analyzed (Participants) | 164 | 147 | 139 | 145 | 140 | 149 | 884
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 164 | 0 | 139 | 0 | 140 | 0 | 443
  >=65 years | 0 | 147 | 0 | 145 | 0 | 149 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (2.8) | 67.6 (2.6) | 60.8 (2.7) | 70.5 (2.0) | 61.0 (2.8) | 70.3 (2.0) | 65.0 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 70 | 87 | 69 | 80 | 78 | 512
  Male | 36 | 77 | 52 | 76 | 60 | 71 | 372
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 7 | 1 | 2 | 2 | 20
  Not Hispanic or Latino | 159 | 144 | 132 | 143 | 138 | 147 | 863
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 5 | 4 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 4 | 18 | 6 | 17 | 8 | 61
  White | 154 | 140 | 114 | 132 | 116 | 138 | 794
  More than one race | 2 | 1 | 4 | 0 | 2 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 164 | 147 | 139 | 145 | 140 | 149 | 884

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Local and Systemic Adverse Events
Description: Participants maintained a memory aid to record daily the occurrence of local injection site reactions and systemic reactions for 8 days after vaccination based on their interference with daily activities for subjective symptoms or quantitative measurement of the reaction. All participants reporting events of any severity (mild, moderate, or severe) are counted. For measured reactions, participants are included if the reaction is >0mm.
Time Frame: Days 0 to Day 7 post vaccination
Population: All participants who received vaccination are included. Data were analyzed regardless of age strata as pre-specified in the study protocol.
Measure: Number; unit: participants
Groups:
- Group IA/B: Pneumococcal Vaccine-naive, Single Injection: Open- label, 13-valent pneumococcal conjugate vaccine (PCV13) given as 0.5 mL intramuscular (IM) injection to vaccine-naive adults ages 55-74.
- Group IIA/B: Previous PPSV23, Single Injection: Open-label, randomized PCV13 given as a 0.5 mL IM injection to adults ages 55-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- Group IIAA/BB: Previous PPSV23, Two Injections: Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to adults ages 55-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
Arm/Group | Group IA/B: Pneumococcal Vaccine-naive, Single Injection | Group IIA/B: Previous PPSV23, Single Injection | Group IIAA/BB: Previous PPSV23, Two Injections
Number analyzed (Participants) | 311 | 284 | 288
participants
  Pain | 148 | 153 | 187
  Tenderness | 213 | 180 | 214
  Redness (measurement) | 40 | 47 | 53
  Swelling | 39 | 49 | 45
  Swelling (measurement) | 39 | 48 | 45
  Elevated oral temperature | 5 | 3 | 7
  Feverishness | 18 | 25 | 29
  Malaise | 53 | 56 | 86
  Headache | 44 | 43 | 63
  Nausea | 13 | 14 | 15
  Chills | 17 | 11 | 26
  New muscle pain | 26 | 26 | 36
  Aggravated muscle pain | 9 | 11 | 21
  New joint pain | 11 | 15 | 16
  Aggravated joint pain | 11 | 15 | 21

2. Primary Outcome: Number of Participants Reporting Unsolicited Vaccine-related Adverse Events.
Description: Association with PCV13 was determined by the investigator and defined as "Related", meaning there was a known temporal relationship, or the event was known to occur in association with study product or with a product in a similar class of study products and no alternate etiology was identified.
Time Frame: Up to Day 28 post vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group IA/B: Pneumococcal Vaccine-naive, Single Injection | Group IIA/B: Previous PPSV23, Single Injection | Group IIAA/BB: Previous PPSV23, Two Injections
Number analyzed (Participants) | 311 | 284 | 288
participants | 19 | 14 | 22

3. Primary Outcome: Number of Participants Reporting Vaccine-related Serious Adverse Events.
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation thereof; was a congenital anomaly/birth defect; or may have jeopardized the participant, or required intervention to prevent one of the outcomes. Association with PCV13 was determined by the investigator and defined as "Related", meaning there was a known temporal relationship, or the event was known to occur in association with study product or with a product in a similar class of study products and no alternate etiology was identified.
Time Frame: Up to Day 180 post vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group IA/B: Pneumococcal Vaccine-naive, Single Injection | Group IIA/B: Previous PPSV23, Single Injection | Group IIAA/BB: Previous PPSV23, Two Injections
Number analyzed (Participants) | 311 | 284 | 288
participants | 0 | 0 | 0

4. Primary Outcome: Geometric Mean Titers of Serotype-specific Opsonophagocytic Antibody (OPA) to 12 Vaccine Serotypes at Days 0 and 28 Post Vaccination.
Description: Blood was collected from all participants at Day 0 and Day 28 after receipt of vaccination. The geometric mean for each group was then assessed by serotype-specific opsonophagocytic antibody (OPA).
Time Frame: Day 0 and Day 28 post vaccination
Population: All participants who received vaccination and had immunology samples obtained within the protocol-defined windows for Days 0, 28, and 180 are included. Three additional subjects were excluded for not meeting eligibility criteria or receipt of a non-study vaccine. Data were analyzed regardless of age strata as pre-specified in the study protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group IA/B: Pneumococcal Vaccine-naive, Single Injection | Group IIA/B: Previous PPSV23, Single Injection | Group IIAA/BB: Previous PPSV23, Two Injections
Number analyzed (Participants) | 307 | 277 | 283
Titer
  Serotype 1, Day 0 | 6.8 [6.0 to 7.7] | 20.9 [16.9 to 25.7] | 20.4 [16.9 to 24.6]
  Serotype 1, Day 28 | 216.0 [177.5 to 262.7] | 75.2 [61.4 to 92.1] | 95.1 [78.6 to 115.0]
  Serotype 4, Day 0 | 20.6 [16.6 to 25.5] | 92.3 [72.2 to 117.9] | 81.3 [63.7 to 103.7]
  Serotype 4, Day 28 | 1808.9 [1570.4 to 2083.5] | 926.6 [787.5 to 1090.3] | 1451.3 [1277.3 to 1649.0]
  Serotype 5, Day 0 | 8.8 [7.6 to 10.2] | 53.0 [41.7 to 67.4] | 36.8 [29.3 to 46.1]
  Serotype 5, Day 28 | 509.8 [416.4 to 624.2] | 287.8 [237.1 to 349.4] | 302.8 [249.5 to 367.5]
  Serotype 6A, Day 0 | 24.1 [19.0 to 30.5] | 47.5 [35.9 to 62.8] | 53.8 [41.1 to 70.5]
  Serotype 6A, Day 28 | 3222.1 [2697.1 to 3849.5] | 2256.7 [1867.1 to 2727.6] | 2903.1 [2364.5 to 3564.5]
  Serotype 6B, Day 0 | 48.8 [37.9 to 62.7] | 106.5 [80.9 to 140.2] | 145.4 [111.1 to 190.4]
  Serotype 6B, Day 28 | 2950.8 [2453.0 to 3549.6] | 1767.8 [1421.2 to 2199.0] | 2562.7 [2095.5 to 3134.0]
  Serotype 7F, Day 0 | 74.6 [57.1 to 97.4] | 284.2 [225.0 to 359.0] | 313.4 [250.1 to 392.8]
  Serotype 7F, Day 28 | 4670.1 [4064.9 to 5365.3] | 1692.4 [1445.1 to 1982.0] | 2144.2 [1870.2 to 2458.4]
  Serotype 9V, Day 0 | 91.1 [71.7 to 115.8] | 210.8 [164.5 to 270.2] | 246.6 [193.3 to 314.5]
  Serotype 9V, Day 28 | 2337.5 [2004.9 to 2725.3] | 1067.5 [895.8 to 1272.2] | 1824.9 [1566.0 to 2126.6]
  Serotype 14, Day 0 | 120.8 [94.1 to 155.0] | 370.5 [288.4 to 476.0] | 452.1 [358.6 to 570.0]
  Serotype 14, Day 28 | 1667.3 [1400.6 to 1984.8] | 1102.2 [916.4 to 1325.7] | 1342.5 [1149.1 to 1568.4]
  Serotype 18C, Day 0 | 41.3 [33.4 to 51.1] | 206.5 [164.0 to 260.0] | 200.8 [157.2 to 256.5]
  Serotype 18C, Day 28 | 2133.1 [1801.8 to 2525.3] | 948.3 [796.1 to 1129.6] | 1373.2 [1181.6 to 1596.0]
  Serotype 19A, Day 0 | 159.2 [131.4 to 193.0] | 540.4 [446.4 to 654.1] | 499.8 [407.9 to 612.4]
  Serotype 19A, Day 28 | 2981.9 [2610.4 to 3406.3] | 1828.8 [1608.6 to 2079.1] | 2316.3 [2046.2 to 2622.1]
  Serotype 19F, Day 0 | 64.8 [52.6 to 80.0] | 153.4 [123.7 to 190.2] | 169.4 [138.8 to 206.6]
  Serotype 19F, Day 28 | 1415.5 [1237.2 to 1619.6] | 727.6 [622.2 to 850.9] | 1050.7 [912.1 to 1210.3]
  Serotype 23F, Day 0 | 17.8 [14.1 to 22.3] | 52.6 [40.7 to 68.0] | 50.6 [39.3 to 65.3]
  Serotype 23F, Day 28 | 947.4 [762.2 to 1177.4] | 652.7 [515.2 to 827.0] | 834.4 [674.5 to 1032.2]

5. Secondary Outcome: Immunogenicity: Serotype-specific OPA Titer to 12 Vaccine Serotypes at Days 0 and 180 Post Vaccination.
Description: Blood was collected from all participants at Days 0 and 180 after receipt of vaccination. The geometric mean for each group was then assessed by serotype-specific opsonophagocytic antibody (OPA).
Time Frame: Day 0 and Day 180 post vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group IA/B: Pneumococcal Vaccine-naive, Single Injection | Group IIA/B: Previous PPSV23, Single Injection | Group IIAA/BB: Previous PPSV23, Two Injections
Number analyzed (Participants) | 307 | 277 | 283
Titer
  Serotype 1, Day 0 | 6.8 [6.0 to 7.7] | 20.9 [16.9 to 25.7] | 20.4 [16.9 to 24.6]
  Serotype 1, Day 180 | 93.4 [76.4 to 141.1] | 45.4 [36.9 to 55.9] | 54.4 [45.1 to 65.7]
  Serotype 4, Day 0 | 20.6 [16.6 to 25.5] | 92.3 [72.2 to 117.9] | 81.3 [63.7 to 103.7]
  Serotype 4, Day 180 | 718.3 [619.4 to 833.1] | 483.9 [407.4 to 574.6] | 734.9 [641.8 to 841.6]
  Serotype 5, Day 0 | 8.8 [7.6 to 10.2] | 53.0 [41.7 to 67.4] | 36.8 [29.3 to 46.1]
  Serotype 5, Day 180 | 234.6 [190.7 to 288.6] | 185.4 [151.6 to 226.8] | 167.6 [136.4 to 205.8]
  Serotype 6A, Day 0 | 24.1 [19.0 to 30.5] | 47.5 [35.9 to 62.8] | 53.8 [41.1 to 70.5]
  Serotype 6A, Day 180 | 1568.5 [1321.6 to 1861.6] | 1155.8 [962.2 to 1388.4] | 1384.4 [1132.5 to 1692.4]
  Serotype 6B, Day 0 | 48.8 [37.9 to 62.7] | 106.5 [80.9 to 140.2] | 145.4 [111.1 to 190.4]
  Serotype 6B, Day 180 | 1425.1 [1188.9 to 1708.2] | 996.1 [806.8 to 1229.9] | 1335.8 [1084.0 to 1646.2]
  Serotype 7F, Day 0 | 74.6 [57.1 to 97.4] | 284.2 [225.0 to 359.0] | 313.4 [250.1 to 392.8]
  Serotype 7F, Day 180 | 2329.0 [2053.3 to 2641.8] | 1063.3 [913.6 to 1237.6] | 1386.9 [1224.5 to 1570.8]
  Serotype 9V, Day 0 | 91.1 [71.7 to 115.8] | 210.8 [164.5 to 270.2] | 246.6 [193.3 to 314.5]
  Serotype 9V, Day 180 | 1191.7 [1016.9 to 1396.5] | 722.4 [602.3 to 866.5] | 1142.8 [979.2 to 1333.7]
  Serotype 14, Day 0 | 120.8 [94.1 to 155.0] | 370.5 [288.4 to 476.0] | 452.1 [358.6 to 570.0]
  Serotype 14, Day 180 | 992.3 [844.3 to 1166.1] | 838.3 [692.2 to 1015.3] | 1056.5 [908.3 to 1229.0]
  Serotype 18C, Day 0 | 41.3 [33.4 to 51.1] | 206.5 [164.0 to 260.0] | 200.8 [157.2 to 256.5]
  Serotype 18C, Day 180 | 964.7 [806.2 to 1154.5] | 590.9 [490.7 to 711.5] | 778.4 [655.0 to 925.2]
  Serotype 19A, Day 0 | 159.2 [131.4 to 193.0] | 540.4 [446.4 to 654.1] | 499.8 [407.9 to 612.4]
  Serotype 19A, Day 180 | 1522.3 [1340.3 to 1728.9] | 1272.1 [1120.7 to 1444.1] | 1508.3 [1326.3 to 1715.3]
  Serotype 19F, Day 0 | 64.8 [52.6 to 80.0] | 153.4 [123.7 to 190.2] | 169.4 [138.8 to 206.6]
  Serotype 19F, Day 180 | 702.3 [612.2 to 805.5] | 481.4 [412.3 to 562.0] | 607.1 [524.9 to 702.2]
  Serotype 23F, Day 0 | 17.8 [14.1 to 22.3] | 52.6 [40.7 to 68.0] | 50.6 [39.3 to 65.3]
  Serotype 23F, Day 180 | 490.7 [394.1 to 611.0] | 353.7 [277.2 to 451.4] | 435.7 [349.2 to 543.5]

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after vaccination, unsolicited AEs through 28 days after vaccination, and SAEs through 180 days after vaccination.
Groups:
- IIA: Previous PPSV23, Age 55-64, Single Injection: Open-label, randomized PCV13 given as a 0.5 mL IM injection to adults ages 55-64 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- IIB: Previous PPSV23, Age 65-74, Single Injection: Open-label, randomized PCV13 given as a 0.5 mL IM injection to adults ages 65-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- IIAA: Previous PPSV23, Age 55-64, Two Injections: Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to adults ages 55-64 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
- IIBB: Previous PPSV23, Age 65-74, Two Injections: Open-label, randomized PCV13 given as a 0.5 mL IM injection in the right arm and 0.5 mL PCV 13 IM in the left arm, to adults ages 65-74 with previous 23-valent pneumococcal polysaccharide vaccine (PPSV23) 3-7 years prior to enrollment.
Arm/Group | IA: Pneumococcal Vaccine-naive, Age 55-64, Single Injection | IB: Pneumococcal Vaccine-naive, Age 65-74, Single Injection | IIA: Previous PPSV23, Age 55-64, Single Injection | IIB: Previous PPSV23, Age 65-74, Single Injection | IIAA: Previous PPSV23, Age 55-64, Two Injections | IIBB: Previous PPSV23, Age 65-74, Two Injections
Serious Adverse Events (participants affected / at risk) | 7/164 | 4/147 | 2/139 | 3/145 | 4/140 | 5/149
Other Adverse Events (participants affected / at risk) | 146/164 | 113/147 | 124/139 | 115/145 | 126/140 | 131/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IA: Pneumococcal Vaccine-naive, Age 55-64, Single Injection (N=164) | IB: Pneumococcal Vaccine-naive, Age 65-74, Single Injection (N=147) | IIA: Previous PPSV23, Age 55-64, Single Injection (N=139) | IIB: Previous PPSV23, Age 65-74, Single Injection (N=145) | IIAA: Previous PPSV23, Age 55-64, Two Injections (N=140) | IIBB: Previous PPSV23, Age 65-74, Two Injections (N=149)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IA: Pneumococcal Vaccine-naive, Age 55-64, Single Injection (N=164) | IB: Pneumococcal Vaccine-naive, Age 65-74, Single Injection (N=147) | IIA: Previous PPSV23, Age 55-64, Single Injection (N=139) | IIB: Previous PPSV23, Age 65-74, Single Injection (N=145) | IIAA: Previous PPSV23, Age 55-64, Two Injections (N=140) | IIBB: Previous PPSV23, Age 65-74, Two Injections (N=149)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 5 (5) | 3 (3) | 11 (11) | 9 (9) | 18 (18)
Vaccination site bruising (General disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 7 (7) | 6 (6)
Feeling hot (General disorders) | 9 (9) | 9 (9) | 17 (17) | 8 (8) | 16 (16) | 13 (13) — Solicited on the memory aid as "Feverishness"
Malaise (General disorders) | 30 (30) | 23 (23) | 30 (30) | 26 (26) | 43 (43) | 43 (43) — Solicited on the memory aid as "Fatigue/Malaise (decreased energy)"
Headache (Nervous system disorders) | 29 (29) | 15 (15) | 25 (25) | 18 (18) | 36 (36) | 27 (27)
Nausea (Gastrointestinal disorders) | 9 (9) | 4 (4) | 11 (11) | 3 (3) | 8 (8) | 7 (7)
Chills (General disorders) | 12 (12) | 5 (5) | 5 (5) | 6 (6) | 13 (13) | 13 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (13) | 15 (15) | 11 (11) | 18 (18) | 18 (18) — Solicited on the memory aid as "New muscle pain (exclusive of the injection site)"
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 5 (5) | 6 (6) | 17 (17) | 4 (4) — Solicited on the memory aid as "Aggravated muscle pain (increase in existing pain, exclusive of the injection site)"
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 10 (10) | 5 (5) | 13 (13) | 3 (3) — Solicited on the memory aid as "New joint pain (arthralgia)"
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 6 (6) | 9 (9) | 16 (16) | 5 (5) — Solicited on the memory aid as "Aggravated joint pain (increase in existing pain)"
Injection site pain (General disorders) | 87 (87) | 61 (61) | 86 (86) | 67 (67) | 94 (94) | 93 (93) — Solicited on the memory aid as "Pain"
Injection site pain (General disorders) | 120 (120) | 93 (93) | 88 (88) | 92 (92) | 109 (109) | 105 (105) — Solicited on the memory aid as "Tenderness"
Injection site erythema (General disorders) | 23 (23) | 17 (17) | 22 (22) | 25 (25) | 31 (31) | 22 (22) — Solicited on the memory aid as "Redness/erythema measurement", reported as experienced if size >0mm
Injection site swelling (General disorders) | 20 (20) | 19 (19) | 24 (24) | 25 (25) | 24 (24) | 21 (21) — Solicited on the memory aid as "Swelling/induration"
Injection site swelling (General disorders) | 21 (21) | 18 (18) | 24 (24) | 24 (24) | 23 (23) | 22 (22) — Solicited on the memory aid as "Swelling/induration measurement", reported as experienced in size >0mm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less